CLINICAL TRIAL: NCT00040300
Title: A 14-Day Study of Racivir When Used in Combination in HIV-Infected Males
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Pharmasset (Industry)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: CI-PSI-004-02-101
Record Dates: First submitted 2002-06-24; First posted 2002-06-25 (Estimated); Last update posted 2005-07-21 (Estimated); Status verified 2005-07

CONDITIONS: HIV Infections
Keywords: treatment experienced; HIV; Phase I; Combination Therapy
MeSH Terms: conditions — HIV Infections | interventions — Racivir

INTERVENTIONS:
Drug: Racivir

SUMMARY:
The purpose of this study is to evaluate Racivir. The safety, most effective dosage, and how the body reacts to Racivir will be studied.

DETAILED DESCRIPTION:
The study is a 14-day study with a 21-day follow-up period. During the 14-days of active study period, participants will receive Racivir once daily in combination with efavirenz and stavudine. Following the administration of the first and last dose of study medication, patients will remain in the clinic overnight. During the study there will be medical and medication histories taken, physical examinations, vital sign measurements, EKGs, and routine clinical laboratory tests.

ELIGIBILITY:
Inclusion Criteria

Subjects may be eligible to participate if they:

* Are males with HIV infection with a positive HIV antibody test
* Have an HIV-RNA copy number of ≥ 5000 copies/ml (Roche assay)
* Have CD4+ cell counts ≥ 50 cells/ml
* Are 18-45 years of age, inclusive
* Have a body mass index (BMI) ≥ 18 kg/m2
* Are antiretroviral nucleoside reverse transcriptase inhibitor-naive
* Have read and understand the informed consent,and is able and willing to comply with study procedures

Exclusion Criteria

Subjects may not participate if they:

* Have clinically significant ECG abnormalities
* Have clinically significant abnormalities in any safety laboratory parameters
* Have an ALT value ≥ 3xUNL
* Have previously participated in this trial
* Have participated in another trial of an investigational drug within the last 3 months or are currently participating in another trial of an investigational drug
* Have a history of chronic alcohol or drug abuse within the last 6 months
* Have a positive urine drug screening
* Have a positive alcohol breath test
* Have any medical or psychiatric condition, which in the opinion of the investigator would jeopardize or compromise the subject's ability to participate in this trial
* Have a known hypersensitivity to any components of the trial medication or comparative drugs as stated in this protocol

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 18
Dates: Start 2002-06; Study Completion 2002-12